CLINICAL TRIAL: NCT01991769
Title: Negative Postprandial Effect on Endothelium After a Not-healthy Meal in Type 2 Diabetes as Affected by Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2011/1801
Record Dates: First submitted 2013-10-28; First posted 2013-11-25 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: exercise; endothelium; postprandial period
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- exercise diabetes type 2 (Experimental): 4x4 min interval training, 47 min moderate intensity training, or no exercise preceding an 'unhealthy' meal.
  Interventions: Behavioral: 47 min moderate intensity training; Behavioral: exercise healthy volunteers; Behavioral: control; no exercise training
- exercise healthy volunteers (Active Comparator): 4x4 min interval training, 47 min moderate intensity training, or no exercise preceding an 'unhealthy' meal.
  Interventions: Behavioral: 47 min moderate intensity training; Behavioral: exercise healthy volunteers; Behavioral: control; no exercise training

INTERVENTIONS:
Behavioral: 47 min moderate intensity training
Behavioral: exercise healthy volunteers
Behavioral: control; no exercise training

SUMMARY:
The purpose of this study is to examine whether exercise reduces the postprandial effects of an unhealthy meal on heart function and endothelial function.

Both healthy people and type 2 diabetes subjects will during three days either carry out two different sessions of exercise training or not before ingesting an unhealthy meal high in saturated fat and fast carbohydrates. The two different exercise training modes used are high intensity interval training (HIIT) and moderate intensity training (MIT) Hypothesis: Exercise training in advance of an unhealthy meal will improve endothelial- and cardiac function in healthy and type 2 diabetes individuals. HIIT will reduce the negative postprandial effects on the endothelium more than MIT.

ELIGIBILITY:
Inclusion Criteria:

* healthy or type 2 diabetes

Exclusion Criteria:

* type 2 diabetes more than 10 years
* unstable angina
* myocardial infarction
* overt cardiovascular disease.
* severe valvular disease.
* overt lung disease.
* orthopedical- /neurological restrictions
* severe disease related to diabetes type 2 (neuropathy, micro-or macroalbuminuria, retinopathy)
* body mass index >35
* severe eating disorders.
* personality disturbances.
* planned surgery during the project period.
* patients who achieve greater than the current exercise guidelines for type 2 diabetes (210 min/week) before the start of the study.
* uncontrolled hypertension
* kidney failure
* cardiomyopathy
* smoking
* patients who probably not will be able to complete the study
* alcohol or drug abuse

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-02; Primary Completion 2012-12 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
endothelial function | 24 hours
  measured as flow mediated dilatation (FMD) of the brachial artery using high resolution vascular ultrasound according to current guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte B Ingul, PhD, Study Director — Norwegian University of Science and Technology
Locations (2):
- Norway (2):
  - Forskningsposten, St Olavs Hospital, Trondheim
  - ISB, Trondheim

REFERENCES:
- [Result] Hollekim-Strand SM, Malmo V, Follestad T, Wisloff U, Ingul CB. Fast food increases postprandial cardiac workload in type 2 diabetes independent of pre-exercise: A pilot study. Nutr J. 2015 Aug 14;14:79. doi: 10.1186/s12937-015-0069-1. PMID 26272328